CLINICAL TRIAL: NCT04812808
Title: Bazedoxifene as a Concomitant Treatment of Patients With Metastatic Pancreatic Adenocarcinoma
Acronym: BAZE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Vignot Lucie, Senior physician, Department of Oncology, Principal Investigator, Hôpital Fribourgeois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Grant-2104
Record Dates: First submitted 2021-03-12; First posted 2021-03-24 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — bazedoxifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bazedoxifene administered in addition to standard chemotherapy protocol (Experimental)
  Interventions: Drug: Bazedoxifene 20 mg

INTERVENTIONS:
Drug: Bazedoxifene 20 mg — Bazedoxifene will be administered during the duration of the study in the experimental arm together with chemotherapy.
  Prophylactic rivaroxaban (Xarelto®) 10 mg per day orally will be added to avoid thromboembolic events.

SUMMARY:
Bazedoxifene, a selective estrogen receptor modulator is thought to have effective anti-tumoral properties for pancreatic cancer via IL-6 pathway (GP130/STAT3) inhibition.

The objective is to measure IL-6 (GP130/STAT3)-pathway modification on metastasis biopsy of patients with metastatic pancreatic adenocarcinoma before and after treatment with bazedoxifene in addition to chemotherapy.

This study is a single-center, prospective, nonrandomized trial.

DETAILED DESCRIPTION:
This study is a single-center, prospective, non-randomized trial. The population studied will consist of 10 patients of both sexes, aged 18 to 85 years, with a newly diagnosed metastatic pancreatic adenocarcinoma who will undergo palliative treatment with standard first line chemotherapy (Gemcitabine +/- Nab-paclitaxel). Diagnosis must be confirmed by biopsy and metastasis must be accessible for percutaneous biopsy using imaging guidance. Further, only patients with an IL-6 (GP130/STAT3)-pathway activity of more than 5% on diagnostic biopsy will be included .

In addition to chemotherapy, patients will receive 20 mg bazedoxifene (Conbriza®) orally per day, subject to good clinical tolerance and in the absence of a biological contraindication.

Patients will receive bazedoxifene once a day at any time, with or without meals. Initiation of treatment will be simultaneous to the initiation of chemotherapy. Bazedoxifene (Conbriza®) will be prescribed and administered for the duration of the study. To minimize the risk of thrombo-embolic events, prophylactic rivaroxaban (Xarelto®) 10 mg orally once per day will be added for the duration of the bazedoxifene (Conbriza®) intake. Pantoprazole 20 mg once per day will be added in selected patients to minimize gastric complications according to the physician's appreciation. Participants will receive bazedoxifene (Conbriza®) and rivaroxaban (Xarelto®) for the entire study duration from a subinvestigator at treatment initiation visit.

Physical examination with vital parameters, laboratory testing (blood count, liver enzymes, creatinine) and tumor marker (CA 19-9) will be conducted in order to determine the baseline prior to the initiation of the treatment. The quality of life using the EORTC core quality of life questionnaire (QLQ-C30) will also be assessed at that point. Furthermore, the IL-6 pathway activity (GP130/STAT3) will be assessed immunohistochemically on metastasis biopsy before administration of bazedoxifene (Conbriza®). The tissue will be obtained by percutaneous biopsy using imaging guidance. A biopsy performed before study inclusion can be used as baseline to avoid a second biopsy.

Study enrollment and follow-up will be performed by the consultant physician at the HFR Fribourg in the department of oncology. The follow-up will be carried out every 3 to 4 weeks and will consist of a physical examination, vital parameters, laboratory testing (blood count, liver enzymes, creatinine, electrolytes) and tumor marker (CA 19-9). Plasma samples will be collected before and after treatment for storage and samples will be analyzed through next generation sequencing NGS. Quality-of-life will be assessed during the follow-ups and drug adherence will be monitored through patient survey.

After 3 months of treatment, the primary endpoint will be assessed. Thoraco-abdominal CT scan or PET-CT will be performed, and a biopsy of metastasis tissue will be repeated (percutaneous under radiological guidance) for immunohistochemical IL-6 pathway activity (GP130/STAT3) analysis. The activity of bazedoxifene (Conbriza®) on inflammatory pathways and tumor progression will be evaluated by comparing the modification in expression of the IL-6 pathway (GP130/STAT3) from baseline.

Patients will be instructed by the investigator to report the occurrence of any adverse event.

The expected duration of the study for each participant will be 12 to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged from 18 to 85,
* Newly diagnosed metastatic pancreatic adenocarcinoma (stage IV according to AJCC)
* Accessible metastasis for percutaneous biopsy using imaging guidance
* IL-6 (GP130/STAT3)-pathway activity of more than 5% on diagnostic biopsy will be included
* Palliative chemotherapy planned,
* Informed Consent as documented by signature (Appendix Informed Consent Form).

Exclusion Criteria:

* No treatment for pancreatic adenocarcinoma,
* Curative treatment of pancreatic adenocarcinoma,
* No accessible metastasis for biopsy,
* Previous thrombo-embolic events,
* Known hypersensibility or allergy to bazedoxifene or one of the Conbriza excipient,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of childbearing potential.
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Inability to give informed consent,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in IL-6/GP-130/STAT3 pathway expression (%) | 3 months
  Assessment of IL-6 (GP130/STAT3) activity by immunohistochemistry on metastasis biopsy before and after treatment with bazedoxifene in addition to chemotherapy.

SECONDARY OUTCOMES:
Carbohydrate-Antigen 19-9 (CA 19-9) in U/ml | every 3 weeks for 3 months
  The change in tumor marker CA 19-9 as a reflection of tumor progression. CA 19-9 will be measured on blood samples collected every 3 to 4 weeks throughout the trial and compared with the baseline prior to treatment initiation.
Change in Quality of life measured by EORTC QLQ-C30 | every 3 weeks for 3 months
  Quality of life using the quality-of-life questionnaire EORTC QLQ-C30. This variable will be measured every 3 to 4 weeks throughout the trial and compared with the baseline prior to treatment initiation. Score ranging from 0 to 100. High scale score represents a higher response level.
Heart rate (bpm) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
Blood pressure (mmHg) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
Oxygen saturation (%) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
weight (kg) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
body temperature (°Celcius) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
liver enzymes (GOT/ASAT in U/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
liver enzymes (GPT/ALAT in U/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
liver enzymes (GGT in U/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
liver enzymes (alkaline phosphatase in U/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
liver enzymes (bilirubine in umol/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
renal parameters (creatinine in umol/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
electrolytes (sodium in mmol/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
electrolytes (potassium in mmol/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
electrolytes (phosphate in mmol/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
electrolytes (calcium in mmol/l) | every 3 weeks for 3 months
  Assess toxicity of bazedoxifene in combination with chemotherapy. Physical examination will be performed and blood samples, including renal and hepatic parameters, will be analyzed every 3 to 4 weeks.
Number of patients with adverse events | every 3 weeks for 3 months
  Assess the number of patients with adverse events (according to CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Vignot, MD, Principal Investigator — Hôpital Fribourgeois
Locations (1):
- HFR Fribourg - cantonal hospital, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No